CLINICAL TRIAL: NCT05668598
Title: Creation of an Ecological Tool Assessing Episodic Memory in Geriatrics: an Adaptation of the Memory Test With Self-Initiated Items (MAI)
Brief Title: Creation of an Ecological Tool Assessing Episodic Memory in Geriatrics
Acronym: ECOTESTGER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier de Lens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022-02; 2022-A02139-34 (Other: ID-RCB)
Record Dates: First submitted 2022-12-09; First posted 2022-12-30 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Memory Disorders; Neurocognitive Disorders
Keywords: GERIATRICS
MeSH Terms: conditions — Memory Disorders; Neurocognitive Disorders

STUDY DESIGN:
Intervention Model Description: Interventional, prospective, Study case-control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Groupe 1 : with neurocognitive disorders (Other): with neurocognitive disorders
  Interventions: Diagnostic Test: ecological MAI test
- Groupe 2 : without neurocognitive disorders (Other): without neurocognitive disorders
  Interventions: Diagnostic Test: ecological MAI test

INTERVENTIONS:
Diagnostic Test: ecological MAI test — Neuropsychological assessment will be realize to determine presence or absence of neurodegenerative disease.
  Study test is ecological MAI.

SUMMARY:
In this study the participants can be recruited via scheduled consultation and external institutions (associations, senior club..). Neuropsychological assessment will be realize to determine presence or absence of neurodegenerative disease.

Study test is ecological MAI. This test are assigned in two groups (with or without neurocognitive disorders).

DETAILED DESCRIPTION:
In this study the participants can be recruited via scheduled consultation and external institutions (associations, senior club..). Neuropsychological assessment will be realize to determine presence or absence of neurodegenerative disease.

Study test is ecological MAI. Participation will be 30 minutes for patients see in case of routine care and 2h30 for those accompanying the patients and participants recruited in external institutions.

Participants are assigned in two groups. Group 1 : with neurocognitive disorders Group 2 : without neurocognitive disorders

Benefits :

For participants without neurodegenerative disorder, study enables to take control early if anomaly will be detected.

The study permit to have cognitive assessment.

Risk : It's possible that participants feel tired. No constraints for participants seen during scheduled consultation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 70 ans
* Person have good locomotion, move independently
* Personne agree to participate

Groupe 1 : 17≤MMSE≤24 (GRECO) Diagnosis of neurodegenerative diseases (major neurocognitive disorders: Alzheimer, mixed dementia, lobar frontotemporal degeneration, vascular dementia).

Groupe 2 : MMSE ≥ à 25 (GRECO) Without neurodegenerative disease

Exclusion Criteria:

* Person with legal protective measures
* Person deprived of liberty
* Mental retardation or MMSE≤ 16
* Understanding verbal disorders
* Visual major disturbances
* Person with disease causing increased fatigue
* Person with psychiatric pathology excepted anxiety disorder or depression with mild episodes.
* Person not covered by French national health insurance

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-08 (Actual); Primary Completion 2026-03-08 (Estimated); Study Completion 2026-03-09 (Estimated)

PRIMARY OUTCOMES:
To compare performance obtaining to overall score remind ecological MAI between older persons with neurocognitive disorders (groupe 1) and older persons without neurocognitive disorders (groupe 2). | day 1
  Overall score remind ecological MAI test (0 to 12) in two groups.

SECONDARY OUTCOMES:
To compare between case and control the various dimensions of episodic memory: temporal component, space component and association component. | day 1
  Spatial component is defined by localisation score. Score (0 to 12)
To compare between case and control the various dimensions of episodic memory: temporal component, space component and association component. | day 1
  Temporal component is defined by temporal dimension.
  Score (0 to 12)
To compare between case and control the various dimensions of episodic memory: temporal component, space component and association component. | day 1
  Association component is defined by binding score.
  Score (0 to 12)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospiralier de Lens, Lens, France

IPD SHARING:
Plan to Share IPD: No